| Division | : | Worldwide Development |
|------------------|---|-------------------------------------|
| Information Type | : | Statistical and Analysis Plan (SAP) |

| Title | : | Statistical and Analysis Plan for Reporting and Analysis Plan for Phase I, Open-Label, Multi-Center Study to Evaluate Safety, Pharmacokinetics and Pharmacodynamics of GSK2798745 after 28 Day Repeat Oral Administration to Adults with Diabetic Macular Edema |
|---|---|---|
| <b>Compound Number</b> | : | GSK2798745 |
| Clinical Study<br>Identifier | : | 212669 |
| <b>Effective Date</b> | : | 21 Jun 2022 |

# **Description:**

The purpose of this SAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 212669.

This SAP will be provided to the study team members to convey the content of the final statistical analysis deliverable.

Details of mock shells for all endpoints are provided in accompanying Shell document and Appendix 11.

Copyright 2022 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

### SAP Author(s):

| Author | |
|--------|----------------------------------------|
| PPD | |
| PPD | Biostatistics (IQVIA, ABDU, Australia) |

### SAP Team Reviews:

SAP Team Review Confirmations (Method: E-mail)



### Clinical Statistics and Clinical Programming Line Approvals:

Clinical Statistics & Clinical Programming Line Approvals (Method: Veeva Vault TMF eSignature)



# **TABLE OF CONTENTS**

| | | PAGE |
|---|---|---|
| 1. | INTRODUCTION | 5 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | 5 |
| | 2.1. Changes to the Protocol Defined Statistical Analysis Plan. | 5 |
| | 2.2. Study Objective(s) Endpoint(s) | |
| | 2.3. Study Design | |
| | 2.4. Statistical Hypotheses / Statistical Analyses | 9 |
| 3. | | |
| | 3.1. Interim Analysis | |
| | 3.2. End of Treatment Period Analysis/Interim Analysis of 28 D | |
| | OCT and CCI | 10 |
| | 3.3. Final Analyses | 10 |
| 4. | | |
| | 4.1. Protocol Deviations | 12 |
| 5. | CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDL | |
| | | 13 |
| | 5.1. Study Treatment & Sub-group Display Descriptors | |
| | 5.2. Baseline Definitions | |
| | 5.5. Other Considerations for Data Analyses and Data Handling Conventions | g<br>13 |
| 0 | | |
| 6. | STUDY POPULATION ANALYSES | |
| 7. | | |
| | 7.1. Adverse Events Analyses | |
| | 7.2. Adverse Events of Special Interest Analyses | |
| | 7.3. Clinical Laboratory Analyses | |
| | 7.4. Other Salety Analyses | 11 |
| 8. | PHARMACOKINETIC ANALYSES | |
| | 8.1. Pharmacokinetic Analyses | |
| | 8.1.1. Pharmacokinetic Analysis For Intensive PK Sam | |
| | 8.1.2. Population of Interest | |
| | 8.1.3. Statistical Analyses / Methods | 19 |
| 9. | | |
| | 9.1. Primary Pharmacodynamic Analyses | |
| | 9.1.1. Endpoint / Variables | |
| | 9.1.2. Summary Measure | |
| | 9.1.4. Strategy for Intercurrent (Post-Randomization) E | |
| | 9.1.5. Statistical Analyses / Methods | |
| | 9.2. Exploratory Pharmacodynamic Analyses | |
| | CCI | |

CCI

| 10. | REFE | RENCES | 24 |
|---|---|---|---|
| 11. | APPEN | NDICES | 25 |
| | 11.1. | Appendix 1: Exclusions from Per Protocol Population | |
| | 11.2. | Appendix 2: Schedule of Activities | |
| | 11.3. | Appendix 3: Assessment Windows | |
| | | 11.3.1. Definitions of Assessment Windows for Analyses | |
| | 11.4. | Appendix 4: Study Phases and Treatment Emergent Adverse | |
| | | Events | 29 |
| | | 11.4.1. Study Phases | 29 |
| | 11.5. | Appendix 5: Data Display Standards & Handling Conventions | 30 |
| | | 11.5.1. Reporting Process | |
| | | 11.5.2. Reporting Standards | |
| | | 11.5.3. Reporting Standards for Pharmacokinetic | 31 |
| | 11.6. | Appendix 6: Derived and Transformed Data | |
| | | 11.6.1. General | 32 |
| | | 11.6.2. Study Population | 32 |
| | | 11.6.3. Pharmacodynamic | |
| | 11.7. | Appendix 7: Reporting Standards for Missing Data | |
| | | 11.7.1. Safety | |
| | | 11.7.2. Premature Withdrawals | |
| | | 11.7.3. Handling of Missing Data | |
| | 11.8. | Appendix 8: Values of Potential Clinical Importance | |
| | | 11.8.1. Laboratory Values | 34 |
| | | 11.8.2. Vital Signs. | |
| | | 11.8.3. ECG | |
| | | 11.8.4 Ophthalmic Examination Values of Potential Clinical | |
| | | Importance | 35 |
| | 11.9. | Appendix 9: Abbreviations & Trademarks | 37 |
| | | 11.9.1. Abbreviations | |
| | | 11.9.2. Trademarks | |
| | 11.10. | Appendix 10: List of Data Displays | |
| | | 11.10.1. Data Display Numbering | 40 |
| | | 11.10.2. Mock Example Shell Referencing | |
| | | 11.10.3. Deliverables | |
| | | 11.10.4. Study Population Tables | |
| | | 11.10.5. Safety Tables | |
| | | 11.10.6. Safety Figures | |
| | | 11.10.7. Pharmacokinetic Tables | |
| | | 11.10.8. Pharmacodynamic Tables | |
| | | 11.10.9. Pharmacodynamic Figures | |
| | | 11.10.10.ICH Listings | |
| | | 11.10.11. Non-ICH Listings. | |
| | 11.11. | Appendix 11: Example Mock Shells for Data Displays | |

### 1. INTRODUCTION

The purpose of this statistical and analysis plan (SAP) is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 212669.

| Protocol Revision Chronology: | | |
|---|---|---|
| Original Document Number: 2019N404030_00 | Dated: 19-Sep-2019 | Version: Original |
| Original Document Number: 2019N404030_01 | Dated: 11-May-2020 | Version: Amendment 01 |
| Original Document Number: 2019N404030_02 | Dated: 28-Oct-2020 | Version: Amendment 02 |
| Original Document Number: TMF-11874499 | Dated: 24-Mar-2021 | Version: Amendment 03 |
| Original Document Number: TMF-14073254 | Dated: 11-NOV-2021 | Version: Amendment 04 |
| Original Document Number: TMF-14377129 | Dated: 2-Feb-2022 | Version: Amendment 05 |

It is noted that GSK terminated this study due to the futility analysis as described in Section 3.1 of this SAP. The SAP details the analysis that is planned based on the sponsor's decision to terminate the study.

### 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Section 9.4.1.2. | Section 9.1.5. Statistical | A repeated measures model |
| Pharmacodynamics (PD) Analysis | Methodology Specification | will allow to model data |
| | | collected at all visits in a |
| A Bayesian probability model will | The primary analysis is | single model and does not |
| be used to analyse the mean | changed to a Bayesian | require an assumption that |
| change from baseline in OCT at | Repeated Measure | the SD is known. |
| Day 28. | Analysis. | |
| Section 9.3 | Section 4 | Site number PPD was closed |
| Populations for Analysis | Analysis Populations | prematurely due to |
| | | significant quality issues. |
| Modified Safety Population has | The modified Safety | Specifically, the following |
| been included in SAP. | Population includes "All | were observed: |
| | subjects in the Safety | |
| | population excluding | <ul> <li>Protocol non-compliance</li> </ul> |
| | subjects from Site number: | <ul> <li>ICF deficiencies</li> </ul> |
| | PPD | <ul> <li>Investigational Product</li> </ul> |
| | | dosing concerns |
| | | <ul> <li>Inadequate source</li> </ul> |
| | | documentation and |
| | | multiple source |
| | | documentation |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| | | deficiencies / inconsistencies • Significant delay in the CRA's access to the Electronic Medical Records (EMR). |
| | | Based on these findings, the site PPD data are considered in question and incomplete. The Analysis Population definitions and resultant Data Displays have been adjusted to address these considerations. |
| | | All safety and relevant study population tables will be undertaken using the Modified Safety Set. Selected safety (Overall and Ocular AE and SAEs) will be repeated for the full safety population. |
| Appendix 10 and 11 | Reductions in the number of tables, listings and figures | Due to study termination due<br>to futility, the number of<br>TFLs being presented has<br>been reduced |
| Section 9 | Bayesian repeated mixed model changed to Bayesian mixed model | Due to termination, analysis will now only consider the baseline and 28 Day visit. Day 14 no longer included in final model |

# 2.2. Study Objective(s) Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary | Primary |
| To characterize the safety and<br>tolerability of GSK2798745<br>following 28 days of daily oral dose<br>administration to adult subjects with<br>confirmed Diabetic Macular Edema<br>(DME). | <ul> <li>Safety parameters including: complete ophthalmic<br/>examination, visual acuity, physical examination findings,<br/>vital sign measurements, clinical lab tests, 12-lead ECG,<br/>clinical monitoring and observation and adverse event<br/>reporting.</li> </ul> |
| <ul> <li>To evaluate the pharmacodynamics<br/>of 28 daily oral doses of<br/>GSK2798745 in the study eye of<br/>adult subjects with DME.</li> </ul> | <ul> <li>Mean change from baseline in center subfield retinal<br/>thickness in the study eye as measured by SD-OCT.</li> </ul> |
| Secondary | Secondary |
| To evaluate the pharmacokinetics<br>of 28 daily oral doses of<br>GSK2798745 in adult subjects with<br>DME. | <ul> <li>Plasma concentrations of GSK2798745, major metabolite<br/>M1, and derived PK parameters, as data permit.</li> </ul> |
| Exploratory | Exploratory |
| CCI | |

## 2.3. Study Design



## 2.4. Statistical Hypotheses / Statistical Analyses

The first co-primary objective of this study is to estimate the treatment effect on mean change from baseline in center subfield retinal thickness in the study eye as measured by SD-OCT at 28 days.

To ensure high probability of accurate decision making around the change at Day 28 in SD-OCT, the decision criteria are defined as:

"Positive" if Prob [CFB in OCT @ 28days > 70 µm decrease|data] > 80% and "Negative" if Prob [CFB in OCT @ 28days < 95 µm decrease|data] > 90%.

If neither Positive nor Negative criterion are meet, an evaluation of the mean change from baseline will be performed. A positive outcome will be concluded if the mean change from baseline in eccluded after completing 28 days of dosing is 3 letters or greater as reviewed in the context of all available PD data.

The second co-primary objective is to evaluate safety of and tolerability of the treatment following 28 days of daily oral dose administration to adult subjects with confirmed DME, hence no formal hypothesis will be tested.

The secondary objective is to evaluate the pharmacokinetics of 28 daily oral doses of GSK2798745 and related M1 metabolite in adult study subjects and derive corresponding PK parameters. Hence, no formal hypothesis will be tested.



### PLANNED ANALYSES

### 3.1. Interim Analysis

After approximately 8 participants completed the Day 28 visit, OCT and data will be analysed on an ongoing basis to assess futility and the study may be terminated early if the futility criteria are met. Additional endpoints may be reviewed as well if necessary. Full details will be provided in the interim analysis charter. The ongoing interim analyses will be the responsibility of GSK Biostatistics.

# 3.2. End of Treatment Period Analysis/Interim Analysis of 28 Day SD-OCT and CC

A preliminary summary of 28-day SD-OCT and based on uncleaned data will be performed after the completion of the following sequential steps:

- A minimum of 20 subjects have completed the 28-day treatment period and provided evaluable assessments of SD-OCT and at baseline and at Day 28.
- The source data of SD-OCT from the Reading Center and eCRF data of Demography, Exposure, Disposition and Protocol Deviation is received as SAS datasets. Data needs to be as clean as possible, since this analysis will be done before final data cleaning and database lock/freeze (DBL/DBF) of the study.

The end-of-treatment interim analysis will be the responsibility of IQVIA Statistics and Programming Functions.

# 3.3. Final Analyses

The final study analyses will be performed after the completion of the following sequential steps:

- All enrolled subjects have completed the study.
- All required database cleaning activities have been completed and final database lock (DBL) has been declared by Data Management.
- 3. The dry runs have been completed prior to the DBL for review by the study team.

These analyses will be the responsibility of IQVIA Statistics and Programming Functions.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All subjects who were screened for eligibility | Screen failures |
| Enrolled | All subjects who passed screening and are<br>eligible for the study with intension to dose. Note screening failures (who never passed | Study populations |
| | screening even if rescreened) and subjects<br>screened but never enrolled into the study are<br>excluded from the Enrolled population as they<br>did not enter the study. | |
| Safety | All enrolled subjects who received at least one dose of study treatment. | <ul> <li>Study Population</li> <li>Selected Safety Tables</li> <li>Population and Safety listings</li> </ul> |
| Modified Safety | All subjects in the Safety population excluding subjects from Site number: PPD | <ul> <li>Selected Study Population </li> <li>Safety Tables</li> <li>Some selected listings repeated </li> </ul> |
| Pharmacodynamic<br>(PD) | All subjects in the modified Safety population<br>who had at least 1 post-baseline non-missing<br>PD assessment. | Pharmacodynamics<br>analysis |
| Pharmacokinetic<br>(PK) | All participants in the modified Safety<br>population for whom a pharmacokinetic<br>sample was obtained and analysed. | Pharmacokinetic analysis |
| Intensive<br>Pharmacokinetic<br>(PK) | All subjects in the modified Safety population who had intensive PK sampling on Day 7 and Day 28 per section 1.3.3 of the protocol. | Intensive Pharmacokinetic analysis |

Note: "Enrolled" means a participant's, or their legally acceptable representative's, agreement to participate in a clinical study following completion of the informed consent process. Potential participants who are screened for the purpose of determining eligibility for the study, but do not participate in the study, are not considered enrolled.

Refer to Appendix 10: List of Data Displays which details the population used for each display.

<sup>\*</sup> This Site Number PPD and serious quality issues, multiple protocol violations and therefore not deemed reliable.

### 4.1. Protocol Deviations

A protocol deviation is any noncompliance with the clinical trial protocol or Good Clinical Practice (GCP). The noncompliance may be either on the part of the subject, the ,zrA, , ity criteria will be considered an enrolment deviation.

Important protocol deviations, including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study.

Exclusion from the analysis sets due to a deviation will be determined programmatically using the criteria described in the table of Analysis populations above. These deviations will not be included in the SDTM dataset but will be programmed in the protocol deviation analysis (ADaM) dataset. This dataset will be the basis for the summaries and listings of protocol deviations.

Data will be reviewed after locking the database and subjects will be assigned to relevant Analysis populations. Suggested population assignments will be sent to GSK for approval before proceeding with the final analysis.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | |
|------------------------------|---------------|
| Data Displays | for Reporting |
| Description | Order in TLF |
| GSK2798745 3.2 mg OD | 1 |

### 5.2. Baseline Definitions

In general, baseline is defined as the last non-missing pre-dose assessment including scheduled and unscheduled visits, unless stated otherwise.

The following specific scenarios will be considered for baseline definition of all ophthalmic examinations including but not restricted to SD-OCT,

- If Day -1 value is not available and a value from any unscheduled visit within 72 hours prior to Day -1 or Day 1 pre-dose is available, then it will be considered as baseline.
- If multiple values are available, for example, on Day -1 as well as any
  unscheduled visit before Day 1 dosing, then latest assessment will be considered
  as baseline.

A missing baseline assessment will not be imputed.

### 5.3. Multicentre Studies

In this multicentre study, unless specified otherwise in specific displays, the data will be presented in an aggregated manner due to small sample size.

# 5.4. Study Eye and Fellow Eye

The central subfield data analysed and provided by a Central Reading Center will be used for the analyses. The CRF data will not be used for reporting. This data is captured as two records per subject per visit one for the right eye and another for the left eye indicated by the Laterality variable. The identification of the Study Eye will be made by the Randomized Laterality variable which specifies whether the study eye is the right or left eye.

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

### **CONFIDENTIAL**

### 

| Section | Component |
|---------|----------------------------------------------------------------|
| 11.1 | Appendix 1: Exclusions from Per Protocol Population |
| 11.2 | Appendix 2: Schedule of Activities |
| 11.3 | Appendix 3: Assessment Windows |
| 11.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 11.6 | Appendix 6: Derived and Transformed Data |
| 11.7 | Appendix 7: Reporting Standards for Missing Data |
| 11.8 | Appendix 8: Values of Potential Clinical Importance |
| 11.9 | Appendix 9: Abbreviations & Trademarks |
| 11.10 | Appendix 10: List of Data Displays |
| 11.11 | Appendix 11: Example Mock Shells for Data Displays |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Enrolled set, unless otherwise specified.

Study population analyses including summaries of subject , disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, exposure and treatment compliance.

Details of the planned displays or mock shells are presented in <u>Appendix 11: Example Mock Shells for Data Displays</u> and accompanying shells document.

### SAFETY ANALYSES

The primary statistical analysis will be to evaluate the safety and tolerability of GSK2798745 following 28 days of daily oral administration to adult subjects with DME. Safety endpoints including adverse events, vital signs (heart rate and blood pressure), clinical laboratory tests,12-lead ECG and CSSRS will be descriptively summarised and listed.

All Safety and relevant study population tables will be presented using the modified Safety analysis population. Overall Adverse Events, Ocular Adverse Events and Serious Adverse Events will be repeated for the Safety Analysis population. Some population tables will be repeated for subjects who received treatment dosing from site# [6] subjects).

All safety and relevant population listings will be presented using the Safety analysis population. Some safety and population listings will be repeated for the modified safety set as presented in the listing of outputs in <a href="Appendix 10">Appendix 10</a>: List of Data Displays, and accompanying shells document.

## 7.1. Adverse Events Analyses

All adverse events starting on or after the first dose of study treatment will be included in the summaries. Adverse events including Serious (SAEs) and events related to study treatment will be summarised descriptively using frequency and percentages overall and by treatment phases (i.e., pre-treatment and on-treatment as defined in Section 11.4.1). On-treatment adverse events include those that occurred in the follow-up phase.

Adverse events will be coded using the standard Medical Dictionary for Regulatory Affairs (MedDRA dictionary). A Standardised MedDRA Query (SMQ) will be used to identify all Ocular, Non-ocular, and COVID-19 AEs.

The incidence of AEs and SAEs (Fatal and Non-Fatal) of COVID-19, COVID-19 AEs leading to study drug discontinuation, COVID-19 AEs leading to study withdrawal, and COVID-19 AEs by severity, will be obtained from standard AE and SAE summaries, without separate outputs due to small sample size.

If >25% participants report ≥1 COVID-19 AE/ SAE, then summaries of onset and duration of the first occurrence of COVID-19 AEs/ SAEs, and of COVID-19 symptoms (from the COVID-19 eCRF page) will be produced, otherwise not.

AEs will be listed by subjects. The details of the planned displays are provided in <u>Appendix 10: List of Data Displays</u>, and accompanying shells document.

# 7.2. Adverse Events of Special Interest Analyses

There are no other Adverse Events of Special Interest defined in the protocol of this study.

# 7.3. Clinical Laboratory Analyses

Laboratory evaluations will be summarised descriptively and listed. The details of the planned displays are in <u>Appendix 10: List of Data Displays</u>, and accompanying shells document.

# 7.4. Other Safety Analyses

Other non-laboratory safety test results including CSSRS, ECGs and vital signs will be summarised descriptively and listed. The details of the planned displays are presented in <u>Appendix 10: List of Data Displays</u>, and accompanying shells document.

### 8. PHARMACOKINETIC ANALYSES

# 8.1. Pharmacokinetic Analyses

Intensive PK sampling in a subset (n 5) of subjects will be undertaken on Day 7 and Day 28 with all subjects providing a trough PK (C<sub>trough</sub>) sample on these 2 days. The Day 7 PK data will be used to ascertain the systemic exposure of the parent drug at the 3.2mg OD is consistent with the predicted exposure (see Table 1 of Protocol).

The plasma concentrations of GSK2798745 and its major metabolite M1 obtained on day 7 and day 28 will be analysed using non-compartmental methods described below. At end of study, all plasma samples (intensive PK Day 7 and Day 28) and trough samples will be analysed using a non-linear mixed effects analysis and is described in the pharmaco-statistical Section 8.1.3. The Population PK analyses using AUC and C<sub>max</sub> will be reported in a separate PK document, outside of the Clinical Study Report (CSR).

## 8.1.1. Pharmacokinetic Analysis For Intensive PK Sampling

Refer to Appendix 5: Data Display Standards & Handling Conventions Derived Pharmacokinetic Parameters.

All non-compartmental pharmacokinetic derivation for the subjects with intensive PK sampling will be conducted by GSK under auspices of Clinical Pharmacology Modelling & Simulation (CPMS). Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin Professional. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the concentration-time data, as data permits. Pharmacokinetic parameters for both parent drug and metabolite M1 will be undertaken.

From the plasma concentration-time data [intensive sampling group], the following pharmacokinetic parameters will be determined for each subject for parent (GSK2798745) and metabolite (M1), if data permits:

| Parameter | Parameter Description |
|---------------------|-----------------------------------------------|
| C <sub>max</sub> | Maximum observed plasma concentration |
| C <sub>trough</sub> | Trough concentration |
| t <sub>max</sub> | Time to C <sub>max</sub> |
| AUC <sub>0-т</sub> | Area under the curve over the dosing interval |

As the trial was terminated, only trough concentrations (C<sub>trough</sub>) for pharmacokinetic analysis will be provided.

### 8.1.2. Population of Interest

The pharmacokinetic analyses (Non-Compartmental) will be based on the PK population, unless otherwise specified.

### 8.1.3. Statistical Analyses / Methods

Statistics and programming will prepare summaries of derived PK parameters provided by the CPMS team, if data permits.

PK concentration data will be loge-transformed and summarised using geometric mean, 95% CI for the geometric mean, SD of loge-transformed data, %CV<sub>b</sub>, and median, min, max of back-transformed data.

Details of the planned displays are provided in <u>Appendix 10: List of Data Displays</u>, and accompanying shells document.

The following PK modelling will be performed by GSK CPMS, if data permits.

### 8.1.3.1. Pharmaco-Statistical Methodology Specification

### **Endpoint / Variables**

All GSK2798745 plasma concentrations at Day 7 and Day 28 including trough samples

# **Model Summary**

Based on the historical population PK model for GSK2798745, a maximum a posteriori probability (MAP) Bayesian estimator based on the limited number of subjects and samples will be applied to derive population PK parameters and associated inter-subject variability taking into account demographic and physiological status of this population. These parameters will then be used in simulations to derive the  $C_{\text{max}}$  and AUC over dosing interval at steady state for each subject.

Internal validation of the population PK model with this population will be undertaken using standard tools such as visual predictive checks and in accordance with the regulatory guidance https://www.fda.gov/media/128793/download .

The PK metrics for GSK2798745 (C<sub>max</sub>, C<sub>trough</sub>, AUC over dosing interval) will be used to assess any relationship with relevant PD parameter.

### 9. PHARMACODYNAMIC ANALYSES

## 9.1. Primary Pharmacodynamic Analyses

The coprimary endpoint of change from baseline in SD-OCT will be analysed using a Bayesian Analysis model.

### 9.1.1. Endpoint / Variables

Change from baseline in center subfield retinal thickness and center point in the study eye as measured by SD-OCT at 28 days.

## 9.1.2. Summary Measure

Mean change from baseline in SD-OCT at day 28.

### 9.1.3. Population of Interest

The primary pharmacodynamics analyses will be based on the Pharmacodynamic population, unless otherwise specified.

## 9.1.4. Strategy for Intercurrent (Post-Randomization) Events

The intercurrent events identified are:

Permanent Discontinuation of the Study Treatment due to any reason Lack of Compliance to Study Treatment

### 9.1.4.1. Permanent Discontinuation of the Study Treatment due to any reason

For the intercurrent event of treatment discontinuation prior to Day 28, a Principal Stratum Strategy will be used for the Primary Estimand, where we are interested to evaluate the treatment effect on subjects who did not permanently discontinue the treatment before 28 days to establish the proof of mechanism of the drug in this Phase 1b study.

Thus, this Principal Stratum of interest will only include subjects who completed the study treatment until Day 28 and provided evaluable data at baseline and on Day 28.

A supplementary analysis using a Hypothetical Strategy will be performed, where we are interested in a hypothetical situation that the treatment discontinuation would not occur. Data from all subjects whether completed treatment until Day 28 or not will be analysed using the same Bayesian Repeated Measures (BRM) analysis as done for the primary analysis.

### 9.1.4.2. Lack of Compliance to Study Treatment

For the intercurrent event of lack of treatment compliance, a Principal Stratum Strategy will be used, where we are interested in subjects who have a high compliance to treatment (defined as 92% of treatment compliance). This principal stratum will include subjects who complete Day 28 with 92% of treatment compliance.

For all other intercurrent events a Treatment Policy Strategy will be considered for the Study eye.

### 9.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in <u>Appendix 10: List of Data Displays</u>, and accompanying shells document.

### 9.1.5.1. Statistical Methodology Specification

### **Endpoint / Variables**

Change from baseline in subfield retinal thickness in the study eye as measured by SD-OCT at 28 days.

Center Subfield retinal thickness is obtained from data provided by Merit CRO. The variables required from the external data (non-CRF collected data) are:

Thickness Sector (thscr c),

laterality (lateral), ). Laterality is to be matched with Study or Fellow Eye.

Criteria of Center subfield thickness reliable (CTRSFTHR = 'Y).

The values of THSCR\_C must be multiplied by 1000 for reporting.

# Bayesian Analysis Model Specification for the Primary Estimand using Principal Stratum Strategy (28 day Completers Analysis)

The mean change from baseline in OCT at Day 28 is assumed to have a t-distribution with (n-1) degrees of freedom.

The variability will be calculated from the observed data.

Evidence of an effect on 28-day OCT will be evaluated based on the posterior probabilities.

### Model Checking & Diagnostics

Not applicable.

### **Model Results Presentation**

Mean change from baseline, its 90% (equal-tailed) credible interval will be reported.

The posterior probabilities that the CFB > 0  $\mu$ m, CFB > 70  $\mu$ m decrease and CFB < 95  $\mu$ m decrease will be reported for Day 28 completers.



# 9.2. Exploratory Pharmacodynamic Analyses





# 10. REFERENCES

GlaxoSmithKline Document Number TMF-14377129: Study Protocol Amendment 05 of 212669, Phase I, Open-Label, Multi-Center Study to Evaluate Safety, Pharmacokinetics and Pharmacodynamics of GSK2798745 after 28 Day Repeat Oral Administration to Adults with Diabetic Macular Edema .

# 11. APPENDICES

# 11.1. Appendix 1: Exclusions from Per Protocol Population

Per protocol population is not defined in this protocol. Important protocol deviations and exclusions from any other analysis population will be listed.

# 11.2. Appendix 2: Schedule of Activities

For a more detailed Schedule of Activities (SoA), please refer to the Section 1.3. Schedule of Activities of the protocol.

| | | | Treatment Period | | | | | Follow- |
|---|---|---|---|---|---|---|---|---|
| Procedure /<br>Study Day: | Visit 1<br>Screening | Visit 2<br>Baseline | Day 1<br>Week 0 | Visit 3<br>Day 7<br>Week 1 | Visit 4<br>Day 14<br>Week 2 | Visit 5<br>Day 28<br>Week 4 | Early<br>Withdrawal<br>(WD) | up<br>Day 56<br>Week 8 |
| Visit Window | -1 to -14 | -3 to -1 | 1 | 6 8 | 13 16 | 27 30 | | 54 - 58 |
| Informed<br>Consent | X | | | | | | | |
| Outpatient<br>Visit | X | X | | X | X | X | X | X |
| Demography | X | | | | | | | |
| Medical History (include substance usage & medication history) | X | X | | | | | | |
| Complete<br>Physical<br>Examination | X | | | | | | X | X |
| Brief<br>Physical<br>Exam | | X | | | X | X | | |
| 12-Lead ECG | X | X | | $X^1$ | X | $\mathbf{X}^{1}$ | X | X |
| Fecal Occult<br>Blood Test<br>(FOBT) | X | | | | | | | |
| Columbia Suicidality Severity Rating Scale (CSSRS) | X | | | X | X | X | X | X |
| Vital Signs | X | X | | X | X | X | X | X |
| Clinical Chemistry, Hematology & UA (including Cardiac Troponin, CPK) | X | X | | X | X | Х | X | X |
| HbA1c | X | | | | | | | |
| FSH /<br>Estradiol | X | | | | | | | |
| Inclusion /<br>Exclusion<br>Criteria | X | | | | | | | |
| Dispense<br>Study<br>Medication | | Х | | | | | | |
| Compliance<br>Check for<br>Study<br>Medication | | | | X | X | X | X | |
| First Day of<br>Study<br>Treatment | | | X | | | | | |

| Dosing in<br>Clinic | | | | X | X | X | | |
|---|---|---|---|---|---|---|---|---|
| PK – Trough<br>Sampling | | | | x | | х | | |
| PK -<br>Intensive<br>Sampling | | | | х | | Х | | |
| Spectral<br>Domain<br>Optical<br>Coherence<br>Tomography<br>(SD-OCT) | x | х | | | x | x | х | х |
| CCI | | | | | | | | |
| General<br>Ophthalmic<br>Exam | x | x | | | | х | x | х |
| CCI | | | | | | | | |
| AE - SAE<br>Assessment | x | x | х | х | х | х | х | x |
| Concomitant<br>Medication | х | х | х | х | х | х | х | х |

# 11.3. Appendix 3: Assessment Windows

# 11.3.1. Definitions of Assessment Windows for Analyses

There will not be multiple assessments for any of the endpoints and therefore assessment windows will not be used for reporting.

Unscheduled visits will be listed and included in the summary of worst case post-baseline assessments only.

Otherwise, only nominal time as per the protocol SoA will be used for all analysis.

# 11.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 11.4.1. Study Phases

Assessments and Adverse Events (AEs) will be classified according to the time of occurrence relative to taking the first dose of the study treatment.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Date ≥ Study Treatment Start Date (including follow-up period) |

NOTE: Pre-treatment AEs will be listed only.

# 11.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before study treatment start date. |
| Concomitant | Any medication or vaccine (including over-the-counter or prescription medicines, some vitamins, and/or herbal supplements), approved by the Investigator, in consultation with the GSK Medical Monitor, that the participant is receiving on or after the start of study treatment. |

**NOTE:** Please refer to 12: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 11.5. Appendix 5: Data Display Standards & Handling Conventions

### 11.5.1. Reporting Process

| Software | |
|---|---|
| SAS 9.4 software | SAS 9.4 software will be used. |
| Reporting Area | |
| SASAppU8_ADC<br>Server | ··· = |
| Analysis Datasets | |
| Source dataset of SD-OCT from the Reading Center will be used for analysis Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1). | |

#### **Generation of RTF Files**

RTF files will be generated for final analysis results

### 11.5.2. Reporting Standards

#### General

Reporting will follow IQVIA SOP CS\_WI\_BS014 Revision 15 standards.

Table specifications are created for each table output to describe the mapping of derived data to the tables. Specifications are considered optional for listings and figures – but the table specification template options (CS\_TP\_BS023 or CS\_TP\_BS024) will be used when creating specifications for listings and tables. Table, figures and listings displays will be used according to CS\_TP\_BS023 shell standards. Where displays are deemed similar to GSK Standards Library (IDSL) by STL, GSK displays will be used instead.

### **Formats**

IQVIA SOP CS\_WI\_BS014 for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.

Numeric data will be reported at the precision collected on the eCRF.

The reported precision from non eCRF sources will follow the IQVIA SOP CS\_TP\_BS023 but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

Reporting for tables, figures and formal statistical analyses:

Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.

The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.

Reporting for Data Listings:

Planned and actual time relative to study drug dosing will be shown in listings. Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

Unscheduled visits will not be included in summary tables and/or figures. But will be included in the summary of worst-case post-baseline results.

All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|--------------------------------|----------------------------------|
| Continuous Data | N, n, mean, sd, median, min, max |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IQVIA SOP CS_TP_BS023 | |

# 11.5.3. Reporting Standards for Pharmacokinetic

Reporting standards for PK data will be based on current CPMS NCA and POP PK guidance documents.

### 11.6. Appendix 6: Derived and Transformed Data

### 11.6.1. General

### Multiple Measurements at One Analysis Time Point

Not Applicable

### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

### 11.6.2. Study Population

### **Treatment Compliance**

Treatment compliance will be calculated based on the formula:

Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \*
Frequency)

- Frequency is 2 for BID and 1 for daily. Treatment compliance could be greater than 100% if there are
  events of overdose. Cumulative compliance (since Day 1) at each visit will be calculated.
- Planned Treatment Duration is defined as 28 days, with potential 8-week opt-in treatment period.

### Extent of Exposure

- Number of days of exposure to study drug will be calculated based on the formula:
  - Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:
  - Cumulative Dose = Sum of (Number of Days x Total Daily Dose)
- If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

### 11.6.3. Pharmacodynamic

#### SD-OCT

### Change from baseline calculation

Change from Baseline = Post-Dose Visit Value - Baseline Value

CC

Other ophthalmology assessments will be summarised only descriptively using similar change from baseline assessments.

# 11.7. Appendix 7: Reporting Standards for Missing Data

# 11.7.1. Safety

| ULN of Laboratory Results |
|--------------------------------------------------------------------|
| Fold Upper Limit of Normal calculation |
| Fold ULN = Laboratory value / the Upper Limit of the Normal range. |

| LLN of Laboratory Results |
|--------------------------------------------------------------------|
| Fold Lower Limit of Normal calculation |
| Fold LLN = Laboratory value / the Lower Limit of the Normal range. |

### 11.7.2. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject's completion is defined as the completion of 28-day treatment period and provide an evaluable assessment of SD-OCT at 28 day Unscheduled assessments will only be included in listings |

# 11.7.3. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table. Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such In this analysis dataset, a missing assessment at any scheduled visit will be considered unevaluable, will not be imputed and will not be included in data analysis. Only observed (OC) cases will be included for all primary, secondary |
| | and exploratory endpoints. |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 11.7.3.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| | Where necessary, display macros may impute dates as temporary variables for |
| | sorting data in listings only. |

# 11.8. Appendix 8: Values of Potential Clinical Importance

# 11.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ <b>44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|-------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T. Bilirubin | µmol/L | High | ≥ 1.5x ULN |
| T. Bilirubin + ALT | µmol/L | High | ≥ 1.5x ULN T. Bilirubin |
| | U/L | | 2x ULN ALT |
| D. Bilirubin | µmol/L | High | ≥ 1.5x ULN |

# 11.8.2. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | 90 | 180 |
| Diastolic Blood Pressure | mmHg | 40 | 120 |
| Heart Rate | bpm | 50 | 120 |

# 11.8.3. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc<br>Interval | msec | > 450 ๗ | |
| Absolute PR<br>Interval | msec | < 110 m | > 220 m |
| Absolute QRS<br>Interval | msec | < 75 m | > <b>110</b> m |
| Change from Baseline | | | |
| Increase from<br>Baseline QTc | msec | > <b>60</b> ៧ | |
| NOTES: 1. Represent standard ECG values of PCI for HV studies | | | |

# 11.8.4 Ophthalmic Examination Values of Potential Clinical Importance

| Ophthalmic Parameter | Potential clinical concern |
|---|---|
| SD-OCT | If a patient has a central subfield change of >120 µm (this corresponds approximately with >15 letter change [Current Opinion in Ophthalmology 2010, 21:172–177]), as assessed by SD-OCT, then this assessment will be categorized as clinically significant. |
| CCI | |
| IOP | If a patient has an IOP assessment which indicates hypo- or hypertonia as follows: Change from baseline of >= 5 mmHG IOP >= 25 mmHG IOP <8 mmHG Increase of >= 5mmHG from previous visit>= 5 mmHg difference between the two eyes at the same visit then this assessment will be categorized as clinically significant. |
| Pupil: pupillary defect | Any post-baseline finding of "Present" Afferent papillary defect (APD) in either eye if APD was not present in that eye at the baseline exam. |
| Motility | Post-baseline changes in eye motility in either eye if motility was normal in that eye at the baseline exam. |

| Ophthalmic Parameter | Potential clinical concern |
|---|---|
| Confrontation visual field | New post-baseline defects in the confrontation visual field. |
| Exam of upper and | Any serious change from baseline by clinical judgment of the investigator |
| lower eyelids | captured as an AE. |
| Meibomian gland | Post-baseline 2-step worsening or 2+ worse per eye. PCIs include: |
| dysfunction | A subject that goes from absent to "obvious inspissation/mild |
| ., | injection, not trichiasis or lid thickening" or "inspissation, debris, obvious |
| | injection, lid thickening, may have trichiasis" |
| | 2) A subject that goes from "mild inspissation/debris without injection or |
| | thickening" to "inspissation, debris, obvious injection, lid thickening, may have |
| | trichiasis" |
| Conjunctival injection or | 2-step worsening and 2+ or worse per eye change from baseline in dilation of |
| chemosis | conjunctival vessels, cilliary injection, subconjunctival hemorrhage, diffuse |
| | edema, subconj. fluid or prolapse of conj. over lower lid. |
| Tear Exam | Any serious change from baseline by clinical judgment of the investigator |
| | captured as an AE. |
| Cornea Epithelium | 2+ worsening change from baseline for edema (i.e., a change from |
| | none to mild patchy microcystic changes), |
| | Any new opacity or whorl-like pattern |
| Corneal Stroma | Any serious change from baseline by clinical judgment of the investigator |
| | captured as an AE. |
| Corneal endothelium | Any serious change from baseline by clinical judgment of the investigator |
| | captured as an AE. |
| Anterior chamber cells | Post-baseline finding of Grade 2+ or worse per eye |
| Anterior chamber | Any post-baseline finding of Present per eye |
| hypopyon | |
| Anterior chamber flare | Any post-baseline finding of Grade 2+ or worse per eye |
| Lens Opacity | 2+ or worse increase in any opacity as compared to baseline per eye (this |
| | can include cortical, nuclear, subcapsular). Any change to "cannot evaluate" |
| | will be flagged as PCI. |
| | The increase will be coloulated by using the following codes: |
| | The increase will be calculated by using the following codes: 1 - <1.0 = no Nuclear/Cortical/any subcapsular opacity, or less than Std. #1 |
| | 2 - 1.0 = Nuclear/Cortical/any subcapsular opacity, or less than std. #1 |
| | 3 - 1.5 = Nuclear/Cortical/any subcapsular opacity between Std. #1 and Std. |
| | #2 |
| | 4 - 2.0 = Nuclear/Cortical/any subcapsular opacity similar to Std. #2 |
| | 5 - 2.5 = Nuclear/Cortical/any subcapsular opacity between Std. #2 and Std. |
| | #3 |
| | 6 - 3.0 = Nuclear/Cortical/any subcapsular opacity similar to Std. #3 |
| | 7 - >3.0 = Nuclear/Cortical/any subcapsular opacity greater than Std. #3 |
| | 8 - 8.0 = cannot evaluate |
| Iris | None |
| Vitreous | Any serious change from baseline by clinical judgement of the investigator |
| | captured as an AE. |
| Optic nerve head | Any serious change from baseline by clinical judgement of the investigator |
| | captured as an AE. |
| Posterior pole | Any serious change from baseline by clinical judgement of the investigator |
| | captured as an AE. |
# 11.9. Appendix 9: Abbreviations & Trademarks

## 11.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| ALT | Alanine aminotransferase (SGPT) |
| ANOVA | Analysis of Variance |
| AST | Aspartate aminotransferase (SGOT) |
| AUC | Area under concentration-time curve |
| AUC(0-τ) | Area under the concentration-time curve over the dosing interval |
| CCI | |
| BMI | Body mass index |
| BP | Blood pressure |
| BPM | Beat Per Minute |
| BRM | Bayesian Repeated Measures |
| CI | Confidence Interval |
| CLr | Renal clearance |
| CL | Systemic clearance of parent drug |
| CL/F | Apparent clearance following oral dosing |
| C <sub>max</sub> | Maximum observed concentration |
| CO2 | Carbon Oioxide |
| CPK | Creatine phosphokinase |
| CPMS | Clinical Pharmacokinetics Modeling & Simulation |
| CPSR | Clinical Pharmacology Study Report |
| CPSSO | Clinical Pharmacology Science & Study Operations |
| eCRF | Electronic Case Report Form |
| CSME | Clinically Significant Macular Edema (CCI |
| CSSRS | Suicidality Severity Rating Scale |
| Ctrough | Pre-dose Trough Concentration measured at end of dosing interval |
| CV | Coefficient of variation |
| DA | Disc Area |
| DBP | Diastolic blood pressure |
| DM | Diabetes Mellitus |
| DME | Diabetic Macular Edema |
| DMPK | Drug Metabolism and Pharmacokinetics |
| DNA | Deoxyribonucleic acid |
| DR | Diabetic Retinopathy |
| ECG | Electrocardiogram |
| CCI | |
| EVA | Electronic Visual Acuity |
| CCI | |
| FDA | Food and Drug Administration |
| CCI | |
| GLP | Good Laboratory Practice |
| GSK | GlaxoSmithKline |

| Abbreviation | Description |
|---|---|
| HbA1c | Glycated Hemoglobin |
| HBsAg | Hepatitis B surface antigen |
| h/hr | Hour(s) |
| HR | Heart rate |
| IB | Investigator's Brochure |
| ICH | International Conference on Harmonization of Technical Requirements for |
| | Registration of Pharmaceuticals for Human Use |
| IDSL | Integrated Data Standards Library |
| IND | Investigational New Drug |
| IP | Investigational Product |
| IRB | Institutional Review Board |
| IU | International Unit |
| IV | Intravenous |
| Kg | Kilogram |
| L | Liter |
| LDL | Low-density lipoprotein |
| LE | Left Eye |
| LFTs | Liver function tests |
| In | Naperian (natural) logarithm |
| LLQ | Lower limit of quantification |
| Lp-PLA2 | Lipoprotein associated phospholipase A2 |
| μg | Microgram |
| μL | Microliter |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Mg | Milligrams |
| mL | Milliliter |
| msec | Milliseconds |
| MMRM | Mixed Models Repeated Measures |
| NCA | Non-Compartmental Analysis |
| NQ | Non-quantifiable concentration measured as below LLQ |
| NVD | New Vessels on Disc |
| NVE | New Vessels – Elsewhere |
| SD-OCT | Optical coherence tomography |
| PA | Preliminary Analysis |
| PC | Phosphatidyl choline |
| PD | Pharmacodynamic |
| PDR | Proliferative Diabetic Retinopathy |
| PGx | Pharmacogenetics |
| рН | Power of Hydrogen |
| PK | Pharmacokinetic |
| PoC | Proof of Concept |
| Pop | Population |
| QC | Quality control |
| RAGE | Receptor for advanced glycation end products |
| RBC | Red blood cells |

| Abbreviation | Description |
|-------------------|--------------------------------------------------|
| RE | Right Eye |
| RNA | Ribonucleic acid |
| SAC | Final Statistical Analysis Complete |
| SAE | Serious adverse event(s) |
| SAP | Statistical and Analysis Plan |
| SAS | Statistical Analysis Software |
| SD | Standard deviation |
| SD-OCT | Spectral domain optical coherence tomography |
| SGOT | Serum glutamic-oxaloacetic transaminase |
| SGPT | Serum glutamic pyruvic transaminase |
| SOP | Standard Operating Procedure |
| SPM | Study Procedures Manual |
| STL | Study Lead Statistician |
| t <sub>1/2</sub> | Apparent Terminal Elimination Half-Life |
| t <sub>last</sub> | Time of last observed quantifiable concentration |
| ULN | Upper limit of normal |
| UK | United Kingdom |
| US | United States |
| VEGF | Vascular Endothelial Growth Factor |
| WBC | White blood cells |

## 11.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| MONOLIX |
| NONMEM |
| RStudio |
| SAS |
| WinNonlin Professional |

### 11.10. Appendix 10: List of Data Displays

Data displays include a combination of displays from standardized GSK IDSL library (with a corresponding reference number as GSK\_XXX), IQVIA specific displays (referenced as IQVIA Tx or IQVIA Lx) and custom, non-standard displays.

A separate document provided the TFL templates is provided with this SAP. These templates describe the presentations for this study and therefore the format and content of the summary tables, figures, and listings to be provided by IQVIA Biostatistics.

### 11.10.1. Data Display Numbering

The following numbering will be applied for SAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|------------|
| Study Population | 1.1 to 1.8 | None |
| Safety | 3.1 to 3.22 | None |
| Pharmacokinetic | 4.1 | None |
| Pharmacodynamic | 6.1 to 6.7 | 6.1 to 6.3 |
| Section | Listi | ngs |
| ICH Listings | 1 to | 13 |
| Other Listings | 14 to | 34 |

#### 11.10.2. Mock Example Shell Referencing

Nonstandard specifications will be referenced as indicated and example mock-up displays provided in <u>Appendix 11: Example Mock Shells for Data Displays</u>, and accompanying shells document.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic | PD_Fn | PD_Tn | PD_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'GSK Statistical Display Standard / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 11.10.3. Deliverables

This section includes deliverables of the IQVIA Statistics and Programming Functions.

| Delivery | Description |
|---|---|
| PA | Preliminary Analysis (also referred to as the End of Treatment Analysis) |
| SAC | Final Statistical Analysis Complete |

# 11.10.4. Study Population Tables

| Study Popu | Study Population Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Shell ID (Output ID) | Title | Programming Notes | Deliverable [Priority] |
| Subject Disposition | | | | | | |
| 1.1. | Screened | GSK_ES6 | GSK_ES6 | Summary of Screening Status<br>and Reasons for Screen<br>Failure | ICH E3 | SAC [1] |
| 1.2. | Safety | GSK_ES1 | GSK_ES1 | Summary of Subject<br>Disposition for the Subject<br>Conclusion Record | ICH E3, Present the data<br>by 2 groups mSafety,<br>Site#PPD | SAC [1] |
| 1.3. | Safety | GSK_SD1 | GSK_SD1 | Summary of Treatment Status<br>and Reasons for<br>Discontinuation of Study<br>Treatment | ICH E3, Present the data by 2 groups mSafety, Site#PPD | SAC [1] |
| Protocol De | eviation | | | | | I |

| Study Popu | Study Population Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Shell ID (Output ID) | Title | Programming Notes Deliverable | |
| 1.4. | Enrolled | GSK_DV1 | GSK_DV1 | Summary of Important<br>Protocol Deviations | ICH E3. Report only the protocol deviations which are defined as important. Present the data by 3 groups Enrolled, msafety and Site#PPD | SAC [1] |
| Population | Analysed | | | | | |
| 1.5. | Enrolled | GSK_SP1 | GSK_SP1 | Summary of Study<br>Populations | | SAC [1] |
| Demograpi | nic and Baseline | Characteristics | | | | |
| 1.6. | Safety | GSK_DM1 | GSK_DM1 | Summary of Demographic<br>Characteristics | ICH E3, FDAAA, EudraCT Present the data by 2 groups mSafety, Site#PPD | SAC [1] |
| 1.7. | mSafety | POP_T1 | POP_T1 | Summary of Diabetes Type by Population | Type 1 and Type 2 | SAC [1] |
| 1.8. | mSafety | GSK_VS1 | DIAB_T1 | Summary of Diabetes<br>Duration | In years | SAC [1] |

# 11.10.5. Safety Tables

| Safety: | Safety: Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Shell ID (Output ID) | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | Adverse Events (AEs) | | | | | |
| 3.1. | Safety | GSK_AE13 | GSK_AE_SUM | Summary of Overall and Ocular Adverse Events | | SAC [1] |
| 3.2. | mSafety | GSK_AE13 | GSK_AE_SUM_mSAF | Summary of Overall and Ocular Adverse Events | | SAC [1] |
| 3.3. | mSafety | IQVIA_T2 | AE007 | Incidence of Ocular and Non-Ocular<br>Adverse Events by System Organ Class<br>and Preferred Term | | SAC [1] |
| 3.4 | mSafety | IQVIA_T2 | AE025 | Incidence of Serious Ocular and Non-<br>Ocular Adverse Events by System Organ<br>Class and Preferred Term | Please display study eye | SAC [1] |
| 3.5 | mSafety | IQVIA_T2 | AE013 | Incidence of Drug-Related Ocular and Non-Ocular Adverse Events by System Organ Class and Preferred Term | and fellow-eye separately as by groups. | SAC [1] |
| 3.6 | mSafety | IQVIA_T2 | AE014 | Incidence of Serious Drug-Related Ocular and Non-Ocular Adverse Events by System Organ Class and Preferred Term | | SAC [1] |
| 3.7 | mSafety | GSK_AE5A | AE019 | Incidence of Ocular and Non-Ocular<br>Adverse Events by System Organ Class<br>and Preferred Term and Maximum<br>Severity | | SAC [1] |

| Safety: | Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Shell ID (Output ID) | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.8 | mSafety | GSK_AE15 | AE030 | Summary of On-Treatment Common (>=x%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC [1] |
| COVID-1 | 19 related AEs | | | | | |
| 3.9 | mSafety | GSK_PAN1 | GSK_PAN1 | Summary of COVID-19 Assessments for Subjects with COVID-19 Adverse Events | | SAC [1] |
| 3.10 | mSafety | GSK_PAN2 | GSK_PAN2 | Summary of COVID-19 Additional<br>Assessments for Subjects with<br>Suspected, Probable or Confirmed<br>COVID-19 Case Diagnosis | | SAC [1] |
| 3.11 | mSafety | IQVIA_PAN1 | IQVIA_PAN1 | Summary of time to onset and duration of first occurrence of COVID-19 Adverse Events | Optional, only if >25% participants reported ≥ 1 COVID-19 AE/SAE | SAC [1] |
| Laborat | ory: Chemistry inc | luding LFT | | | | |
| 3.12 | mSafety | GSK_LB1 | Chem001 | Summary of Chemistry including Liver Function Test Changes from Baseline | Include LFT parameters | SAC [1] |
| 3.13 | mSafety | GSK_LB17 | Chem002 | Summary of Worst-Case Chemistry including Liver Function Test Results by PCI Criteria Post-Baseline Relative to Baseline | Include LFT parameters | SAC [1] |

| Safety: | Safety: Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Shell ID (Output ID) | Title | Programming Notes | Deliverable<br>[Priority] |
| Laborat | ory: Hematology | | | | • | |
| 3.14 | mSafety | GSK_LB1 | Hem001 | Summary of Hematology Changes from Baseline | | SAC [1] |
| 3.15 | mSafety | GSK_LB17 | Hem002 | Summary of Worst-Case Hematology<br>Results by PCI Criteria | | SAC [1] |
| | | | | Post-Baseline Relative to Baseline | | |
| Laborat | ory: Urinalysis | | | | | |
| 3.16 | mSafety | GSK_UR1 | UR001 | Summary of Worst Case Urinalysis Results Post-Baseline Relative to Baseline | | SAC [1] |
| ECG | | | | | | |
| 3.17 | mSafety | IQVIA_T10 | EG001 | Summary of ECG Values and Change from Baseline | | SAC [1] |
| 3.18 | mSafety | IQVIA_T11 | EG002 | Summary of Shift from Baseline in ECG Findings | | SAC [1] |
| Vital Sig | ıns | | | | | |
| 3.19 | mSafety | IQVIA_T10 | VS001 | Summary of Vital Signs Values and Change from Baseline Findings | | SAC [1] |
| 3.20 | mSafety | IQVIA_T13 | VS002 | Summary of Subjects with Vital Sign<br>Results outside PCI Ranges | | SAC [1] |

| Safety: Tables | | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Shell ID (Output ID) | Title | Programming Notes | Deliverable<br>[Priority] |
| Columbia Suicidality Severity Rating Scale (CSSRS) | | | | | | |
| 3.21 | mSafety | GSK_CSSRS1 | CSSR01 | Summary of Subjects with C-SSRS<br>Suicidal Ideation or Behaviour during<br>Treatment | | SAC [1] |
| 3.22 | mSafety | GSK_CSSRS3 | CSSR02 | Shift Table of Changes in C-SSRS<br>Categories from Pre-Treatment to On-<br>Treatment | | SAC [1] |
| 3.23 | mSafety | IQVIA_T13 | EG003 | Summary of Subjects with ECG Results outside PIC Ranges | | SAC [1] |

### CONFIDENTIAL

212669

# 11.10.6. Safety Figures

Not planned due to small sample size.

## 11.10.7. Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. Population GSK Standard / Example Shell ID (Output ID) Title Programming Notes Programming Notes [Priority] | | | | | |
| GSK2798745 ar | GSK2798745 and M1 Metabolite | | | | |
| 4.1. | PK | GSK_PK01 | PK001 | Summary of GSK2798745 and M1 metabolite Pharmacokinetic Concentration-Time Data | SAC [1] |

# 11.10.8. Pharmacodynamic Tables

| No. | Population | GSK<br>Standard/<br>Example Shell | Shell ID<br>(Output ID) | Title | Programming Notes | Deliverable [Priority |
|---|---|---|---|---|---|---|
| SD-OC | D-OCT | | | | | |
| 6.1. | PD | PD_T1 | PD001 | Summary of Center Subfield Retinal<br>Thickness in the Study and Fellow-Eye as<br>Measured by SD-OCT, including change<br>from baseline. | Present study eye and fellow eye as separate by groups | PA, SAC [1] |
| 6.2. | PD | PD_T2 | PD002 | Bayesian Analysis of Change from<br>Baseline in Center Subfield Retinal<br>Thickness in the Study and Fellow Eye as<br>Measured by SD-OCT at Day 28 (Day 28<br>Completers Analysis) | Includes only subjects who have completed Day 28 | PA, SAC [1] |
| CCI | | | | | | |

| Pharma | Pharmacodynamic: Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK<br>Standard/<br>Example Shell | Shell ID<br>(Output ID) | Title | Programming Notes | Deliverable [Priority] |
| CCI | | | | | | |
| - | | | | | | |

| Pharm | Pharmacodynamic: Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK<br>Standard/<br>Example Shell | Shell ID<br>(Output ID) | Title | Programming Notes | Deliverable [Priority] |
| Other | Other Exploratory Endpoints | | | | | |
| CCI | | | | | | |

# 11.10.9. Pharmacodynamic Figures

| Pharmaco | odynamic: Fig | ures | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK<br>Standard/<br>Example Shell | Shell ID (Output ID) | Title | Programming Notes | Deliverable [Priority] |
| SD-OCT | | | | | | |
| | | | | | Mock shell provided is an<br>example figure, not study<br>specific | |
| 6.1. | PD | SAFE_F2 | PDFIG001 | Individual Plot of Change from<br>Baseline in Center Subfield Retinal<br>Thickness in the Study Eye as<br>Measured by SD-OCT | X-axis is visit, Y-axis is change from baseline in center subfield retinal thickness. | PA, SAC [1] |
| | | | | | General comment: Format the intervals based on the interval of time. | |
| CCI | | | | | | |

| No. | Population | GSK<br>Standard/<br>Example Shell | Shell ID (Output<br>ID) | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|---|
| SD-OCT & CCI | | | | | | |
| 6.3. | PD | SAFE_F2 | PDFIG011 | Correlation Plot of Change from Baseline in OCT versus CCI at Day 28. | Mock shell provided is an example figure, not study specific. X-axis is CFB of CCI at Day 28, Y-axis is CFV of SDOCT at Day 28. Also present Pearson's Correlation coefficient (r). | SAC [1] |

# 11.10.10. ICH Listings

| ICH: Lis | ICH: Listings | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Shell ID (Output<br>ID) | Title | Programming Notes | Deliverable [Priority] |
| Subject | Subject Disposition | | | | | |
| 1. | Screened | GSK_ES2 | GSK_ES2 | Listing of Reasons for Study<br>Withdrawal | ICH E3 | SAC [1] |
| 2. | Safety | GSK_SD2 | GSK_SD2 | Listing of Reasons for Study<br>Treatment Discontinuation | ICH E3 | SAC [1] |
| Protoco | ol Deviations | | | | | |
| 3. | Enrolled | GSK_DV2 | GSK_DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC [1] |
| 4. | Enrolled | GSK_IE3 | GSK_IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC [1] |
| Populat | tions Analysed | d | | | | |
| 5. | Enrolled | GSK_SP3 | GSK_SP3 | Listing of Subjects Excluded from Any Population | ICH E3 | SAC [1] |
| Demog | raphic and Ba | seline Characteristics | 3 | | | |
| 6. | Safety | GSK_DM2 | DEMO | Listing of Demographic Characteristics | ICH E3 | SAC [1] |
| 7. | Safety | GSK_DM9 | RACE | Listing of Race | ICH E3. Use Geographic ancestry data. | SAC [1] |
| Exposu | re and Treatm | ent Compliance | | | | |

| ICH: Lis | stings | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Shell ID (Output<br>ID) | Title | Programming Notes | Deliverable [Priority] |
| 8. | Safety | GSK_EX3 | Exposure | Listing of Exposure | ICH E3 | SAC [1] |
| 9.1 | Safety | GSK_COMP2a | Compliance | Listing of Compliance | ICH E3 | SAC [1] |
| 9.2 | Safety | GSK_COMP2a | Noncompl_Reason | Listing of Reasons for Non-<br>Compliance | ICH E3 | SAC [1] |
| Advers | Adverse Events | | | | | |
| 10. | Safety | GSK_AE8 | AEList1 | Listing of All Adverse Events | ICH E3; | PA, SAC [1] |
| 11. | Safety | GSK_AE8 | AEList3 | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | ICH E3 | SAC [1] |
| Serious | Adverse Eve | nts | | | | |
| 12. | Safety | GSK_AE8 | AEList5 | Listing of Serious Adverse<br>Events | ICH E3 | SAC [1] |
| All Lab | oratory | | | | • | |
| 13. | Safety | IQVIA_L1/<br>GSK_LB5 | LABList | Listing of All Laboratory Data<br>for Subjects including Any<br>Value of Potential Clinical<br>Importance | ICH E3; include LFT and Urinalysis parameters | SAC [1] |

# 11.10.11. Non-ICH Listings

| Non-ICH: Listin | ngs | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display<br>Standard / Example<br>Shell | Shell ID (Output ID) | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject Disposition | | | | | | |
| 14 | Screened | GSK_ES7 | SCRFail | Listing of Reasons for<br>Screen Failure | Journal Guidelines | SAC [1] |
| Prior and Cond | comitant Medications | | | • | | |
| 15 | Safety | GSK_CM3 | PM1 | Listing of Diabetes<br>Information | Listing-Other; Including Diabetes type, length of duration (in years) | SAC [1] |
| 16 | Safety | GSK_CM3 | MH1 | Listing of Medical<br>History | | SAC [1] |
| 17 | Safety | GSK_CM3 | PM2 | Listing of Prior<br>Medication by Generic<br>Term | For prior, including a column of relative time to first dosing day (Day 1) (in months, if month is missing, use December); DME medication <sup>4</sup> Listing-Other | SAC [1] |
| 18 | Safety | GSK_CM3 | CM1 | Listing of Concomitant<br>Medication by Generic<br>Term | , , | SAC [1] |
| 19 | Safety | NA | LASERLIST | Listing of Laser History | | SAC [1] |
| Adverse Event | s | | | | | |
| 20 | Safety | GSK_PAN7 | COVList | Listing of All Subjects with Visits or Assessments | | SAC [1] |

| Non-ICH: Listin | ngs | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display<br>Standard / Example<br>Shell | Shell ID (Output ID) | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | | Impacted by COVID-<br>19 | | |
| Hepatobiliary ( | Liver) | | | | | |
| 21 | Safety | IQVIA_L2 | LFTList | Listing of Fold ULN for LFTs | | SAC [1] |
| Ophthalmologi | ical Assessments | | | | | |
| 22 | PD | SAFE_T2 | OPT001 | Listing of General Ophthalmic Examinations Data including Abnormalities of Potential Clinical Importance | Include all subjects in the listing excluding SD-OCT and excluding and flag any values of potential clinical importance | SAC [1] |
| 23 | PD | SAFE_T3 | OPT002 | Listing of Absolute and<br>Change from baseline<br>in SD-OCT Numeric<br>Endpoints for both<br>eyes including<br>Abnormalities of<br>Potential Clinical<br>Importance | Include all subjects in the<br>listing and flag any values of<br>potential clinical importance | SAC [1] |
| 24 | PD | SAFE_T4 | OPT003 | Listing of SD-OCT<br>Non-numeric<br>Endpoints for both<br>eyes including | Include all subjects in the listing and flag any values of potential clinical importance | SAC [1] |

| Non-ICH: Listings | | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display<br>Standard / Example<br>Shell | Shell ID (Output ID) | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | | Abnormalities of<br>Potential Clinical<br>Importance | | |
| 25 | PD | SAFE_T3 | OPT004 | Listing of Absolute and Change from Baseline in Colomb Numeric Endpoints for Study and Fellow Eyes including Abnormalities of Potential Clinical Importance | Include all subjects in the<br>listing and flag any values of<br>potential clinical importance | SAC [1] |
| 26 | PD | SAFE_T4 | OPT005 | Listing of Columnon Non-<br>numeric Endpoints for<br>both eyes included<br>Abnormlities of<br>Potential Clinical<br>Importance | Include all subjects in the<br>listing and flag any values of<br>potential clinical importance | SAC [1] |
| 27 | PD | SAFE_T3 | OPT006 | Listing of Absolute and Change from baseline in Coll and Endpoints for both eyes including Abnormalities of Potential Clinical Importance | Include all subjects in the<br>listing and flag any values of<br>potential clinical importance | SAC [1] |

| Non-ICH: Listin | Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display<br>Standard / Example<br>Shell | Shell ID (Output ID) | Title | Programming Notes | Deliverable<br>[Priority] |
| 28 | PD | SAFE_T4 | OPT007 | Listing of CCI and CCI Non-numeric Endpoints for both eyes including Abnormalities of Potential Clinical Importance | | SAC [1] |
| ECG | | | | | | |
| 29 | Safety | IQVIA_L3 | ECGLIST01 | Listing of Individual 12-<br>lead ECG Results<br>including Any Value of<br>Potential Clinical<br>Importance | | SAC [1] |
| 30 | Safety | GSK_EG5 | ECGLIST02 | Listing of All ECG<br>Findings for Subjects<br>with an Abnormal<br>Finding | | |
| Vital Signs | | | | | | |
| 31 | Safety | IQVIA_L5 | VSLIST01 | Listing of Individual<br>Vital Signs Results<br>including Any Value of<br>Potential Clinical<br>Importance | | SAC [1] |

| Non-ICH: Listings | | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display<br>Standard / Example<br>Shell | Shell ID (Output ID) | Title | Programming Notes | Deliverable<br>[Priority] |
| Columbia Suicidality Severity Rating Scale (CSSRS) | | | | | | |
| 32 | Safety | GSK_CSSRS4 | CSSRLIST01 | Listing of C-SSRS<br>Suicidal Ideation and<br>Behaviour Data | | SAC [1] |
| PK Endpoints | | | | | | |
| 33 | PK | GSK_PK07 | PKLIST001 | Listing of GSK279845<br>and M1 Metabolite<br>Plasma<br>Pharmacokinetic<br>Concentration-Time<br>Data [intensive &<br>C <sub>trough</sub> samples] | | SAC [1] |
| 34 | PK | GSK_PK13 | PKLIST002 | Listing of Derived<br>GSK279845 and M1<br>Metabolite Plasma<br>Pharmacokinetic<br>Paramaters [intensive<br>& Ctrough samples] | | SAC [1] |

# 11.11. Appendix 11: Example Mock Shells for Data Displays

Please refer to the mock shells document.